CLINICAL TRIAL: NCT05663320
Title: A Feasibility Pilot Study of a Virtual Education-Based Transition Intervention to Improve Transition Readiness in Adolescent and Young Adults With Congenital Adrenal Hyperplasia.
Brief Title: A Study of a Virtual Education-Based Transition Intervention to Improve Transition Readiness in Adolescent and Young Adults With Congenital Adrenal Hyperplasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never opened; deemed duplicative of another active NIH protocol.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10000411; 000411-CC
Record Dates: First submitted 2022-12-22; First posted 2022-12-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Self-Paced; Interactive; Adrenal Biomarkers; Trxansition Index Score; Health Care Transition
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Other): Intervention Study Arm 1 participants will receive an approximately 11minute educational video on CAH that focuses on transitional goals (at baseline, 3 months, and 6 months. This will be done via a NIH approved webbased REDCap. Completion will be recorded.
  Interventions: Other: virtual educational based transition intervention self-paced
- 2 (No Intervention): Usual care Study Arm 2 participants will have their usual six-month CAH follow up to coincide with study visits at 0, 6 and 12 months. During their visit, study participants will receive standard care that includes self-injection teaching and sick day rules

INTERVENTIONS:
Other: virtual educational based transition intervention self-paced — study intervention is a standardized, virtual educational video on CAH that will be delivered self-paced
  Arms: 1

SUMMARY:
Background:

Children with congenital adrenal hyperplasia (CAH) can survive well into adulthood with proper treatment. But the change from pediatric to adult care can be challenging. Many people with CAH need extra support as they learn to take control of their own health care needs. Researchers have studied how people respond to different types of patient education. Now researchers want to find out if virtual education, via computer, is a good way to teach people how to manage CAH as they become adults.

Objective:

To test a virtual method of delivering patient education to adolescents and young adults with CAH.

Eligibility:

Adolescents and young adults aged 16 to 22 years who have CAH. They must already be enrolled in Natural History Study Protocol 06-CH-0011.

Design:

Participants may take part in the study remotely; they may also come to the clinic. They will have 3 visits in 1 year.

Participants will complete questionnaires. Topics will include what they know about CAH; whether they remember to take their medications on their own; and whether they schedule their own appointments. They will be asked about their quality of life. They will be asked about their physical and emotional health.

All participants will be taught how to care for themselves. The participants will be divided into 2 groups. Some will watch an 11-minute video on CAH that focuses on their goals as they become adults. The others will receive standard education.

After 6 months, participants will receive CAH education again.

After 12 months, participants will repeat the questionnaires from their first visit.

DETAILED DESCRIPTION:
Study Description:

Health Care Transition (HCT) is defined as planned movement of chronically ill youth and young adults from a child to an adult model of care. HCT initiatives aim to facilitate the transition process and reduce commonly observed complications associated with poor transition such as decreased health literacy, poor treatment adherence, discontinuity of care and poor medical outcomes. The NIH Clinical Center is a unique environment where children with rare diseases such as Congenital Adrenal Hyperplasia (CAH) are often followed longitudinally into adulthood. Rare diseases are understudied and few studies have investigated effective ways of delivering HCT focused education to improve transition readiness. This is a pilot, randomized controlled trial that will assess the feasibility and preliminary efficacy of a virtual education-based transition intervention to improve transition readiness in adolescents and young adults with CAH. We hypothesize that the virtual education-based transition intervention will be feasible and participants in the intervention arm, will have better transition readiness score, disease outcomes and quality of life as compared to participants who received usual care.

Objectives:

Primary objective: To assess the feasibility of a virtual education based transition intervention in adolescents and young adults with CAH.

Secondary Objective: To assess preliminary effectiveness of a virtual education-based transition intervention on measures of transition readiness.

Endpoints:

Primary Endpoint: a) study participant compliance rate of >= 67% with virtual education-based transition intervention, and b) feasibility of collecting all study questionnaires from >=75% of participants at all time periods.

Secondary Endpoint: The change in baseline to 12 months in the University of North Carolina (UNC) Trxansition Index score.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed assent or consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Patients between ages 16-22
* Diagnosed with CAH and enrolled in the Natural History Study Protocol 06-CH-0011.
* Ability to speak and comprehend English as this is a pilot study and the study intervention education video is currently only in English and requires validation before translation into other languages
* Access to a computer/mobile device and the internet.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients with significant medical or cognitive impairment(s) that may interfere with participating in trial.
* Participants unable to participate in all aspects of this clinical trial.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-09 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
UNC Trxansition Index measure | 12 months
  The UNC Trxansition Index is a validated, provider-administered transition readiness questionnaire.

SECONDARY OUTCOMES:
Disease-specific knowledge | 12 months
  Disease-specific knowledge
Self-Management and Transition to Adulthood with Rx (STARx) questionnaire | 12 months
  Self-Management and Transition to Adulthood with Rx (STARx) questionnaire
Degree of disease control based on two commonly used adrenal biomarkers | 12 months
  Degree of disease control based on two commonly used adrenal biomarkers
HRQoL based on Short Form Health Survey (SF-36). | 12 months
  HRQoL based on Short Form Health Survey (SF-36).
Number of hospitalizations per year related to CAH | 12 months
  Number of hospitalizations per year related to CAH
Number of school/work absences per year related to CAH | 12 months
  Number of school/work absences per year related to CAH

CONTACTS AND LOCATIONS:
Overall Officials: Ruth W Parker, C.R.N.P., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000411-CC.html